CLINICAL TRIAL: NCT04120103
Title: Effect of Doll Therapy on the Cognitive States and Agitation Levels of Patients With Moderate and Severe Dementia
Brief Title: Doll Therapy on Patients With Moderate and Severe Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Cemile KÜTMEÇ YILMAZ, Principal Investigator, Aksaray University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017/81
Record Dates: First submitted 2019-08-01; First posted 2019-10-09 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Dementia
Keywords: Dementia; Agitation; Cognitive status; Doll therapy
MeSH Terms: conditions — Dementia; Psychomotor Agitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Doll therapy (Experimental): Experimental: Doll Therapy Intervention A total of 30 patients were included in the study. All patients that meet the study inclusion criteria will be included in the study The patients in the intervention group will have Doll therapy for 60 days and weekly patient visits. The study will be started with control group patients. At the beginning of the study and after 60 days, "Introductory Information Form", Mini Standard Mini Mental Test "and" Cohen-Mansfield Agitation Inventory "will be applied to patients in intervention and control groups for data collection. Dementia patients will be given a baby, patients will be followed for two months. There will be monitoring once a week.
  Interventions: Behavioral: Doll therapy
- Routine nursing care (Active Comparator): The nursing care provided by the institution was applied to the dementia patients in the routine nursing care group. Routine nursing care group interventions in the institution; Monitoring of life signs, application of drug treatments, participation in social activities such as listening to music, reading prayer, initiatives such as assisting patients in performing daily living activities.
  There was no intervention other than routine care. The patients were followed up for two months.The patients were followed up for two months.Data collection forms were applied at the beginning, first and second months of the study.
  Interventions: Other: Routine nursing care

INTERVENTIONS:
Behavioral: Doll therapy — The patient will then be given the doll to be used in the research by the caregiver and the researcher. Intervention group (accepting the baby) will be evaluated in terms of interaction with the baby, communication with employees and other patients and participation in daily life activities for 60 days. In addition, the agitation symptoms of the patients during the 60 days they spend with the baby will be evaluated by CMAI and cognitive level by MMSE.
  Arms: Doll therapy
Other: Routine nursing care — The nursing care provided by the institution was applied to the dementia patients in the routine nursing care group. Routine nursing care group interventions in the institution; Monitoring of life signs, application of drug treatments, participation in social activities such as listening to music, reading prayer, initiatives such as assisting patients in performing daily living activities.
  Arms: Routine nursing care

SUMMARY:
Doll therapy is one of the non-pharmacological methods that can be practiced in managing the symptoms of dementia patients. Nurses can practice doll therapy independently, and literature reports that it has positive effects on the behaviors, moods, emotions, cognitive states and social life of patients with moderate and severe dementia. Our country had no study that investigated the effect of doll therapy in managing the cognitive and behavioral symptoms of dementia patients. This project is a randomized controlled trial that aims to investigate the effect of Doll therapy on the cognitive states and agitation levels of patients with moderate and severe dementia.

DETAILED DESCRIPTION:
Dementia is a progressive neurodegenerative disease increasing in prevalence due to the aging population that grows in parallel with the increased life expectancy at birth in recent years. It is characterized with a progressive deterioration in cognitive abilities and memory. Due to the increasing losses in cognitive and physical functions, people with dementia become in need of nursing over time. Agitation is the most common behavioral symptom.

Agitation is defined as improper verbal, vocal and motor activity that are not purposeful and are not caused by confusion. Verbal and physical aggression, restlessness, aimless wandering, profanity, self-harm, continuous and repetitive questioning behavior emerges.Agitation should be managed with reliable and tolerable, effective methods in order to affect the quality of life of both the patient and the caregiver negatively.

Doll therapy is one of the non-pharmacological methods that can be practiced in managing the symptoms of dementia patients. Nurses can practice doll therapy independently, and literature reports that it has positive effects on the behaviors, moods, emotions, cognitive states and social life of patients with moderate and severe dementia.Our country had no study that investigated the effect of doll therapy in managing the cognitive and behavioral symptoms of dementia patients. This study is a randomized controlled trial that aims to investigate the effect of Doll therapy on the cognitive states and agitation levels of patients with moderate and severe dementia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with moderate to severe dementia (those with a SMMT score of 17 or less)
* Having dexterity to hold or caress a baby
* No problem with communication obstruction
* Dementia patients who agree to participate in the study

Exclusion Criteria:

* Mild stage dementia,
* Diagnosed with neurological or psychiatric diseases other than dementia, not accepting the baby despite two attempts,
* Rarely agitated dementia patients with baby dolls

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Standardized Mini Mental Test | 2 months after the beginning intervention.
  cognitive status
Cohen-Mansfield Agitation Inventory | 2 months after the beginning intervention
  Cognitive and agitation status

CONTACTS AND LOCATIONS:
Overall Officials: Cemile KÜTMEÇ YILMAZ, Dr, Principal Investigator — Aksaray University, Faculty of Health Science, Nursing Department, Turkey
Locations (1):
- Cemile KÜTMEÇ YILMAZ, Merkez, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yilmaz CK, Asiret GD. The Effect of Doll Therapy on Agitation and Cognitive State in Institutionalized Patients With Moderate-to-Severe Dementia: A Randomized Controlled Study. J Geriatr Psychiatry Neurol. 2021 Sep;34(5):370-377. doi: 10.1177/0891988720933353. Epub 2020 Jun 17. PMID 32552299